CLINICAL TRIAL: NCT06803654
Title: A Randomized, Multicenter, Double-Masked, Active-Controlled, Parallel-Group Study Comparing the Efficacy and Safety of Brimonidine Tartrate Ophthalmic Solution 0.025% With Sodium Hyaluronate Relative to Lumify in Adult Subjects With Ocular Redness
Brief Title: A Study Comparing the Efficacy and Safety of Brimonidine Tartrate Ophthalmic Solution 0.025% With Sodium Hyaluronate Relative to Lumify in Adult Subjects With Ocular Redness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BL-CO01-LUMHA-1301
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Ocular Redness
MeSH Terms: interventions — Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant
Masking Description: Double masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brimonidine tartrate ophthalmic solution 0.025% with sodium hyaluronate (BTOS-HA) (Experimental)
  Interventions: Drug: BTOS-HA
- Brimonidine tartrate ophthalmic solution 0.025% (Active Comparator)
  Interventions: Drug: Lumify®

INTERVENTIONS:
Drug: BTOS-HA — Brimonidine tartrate ophthalmic solution 0.025% with sodium hyaluronate (BTOS-HA) administered as 1 topical ocular drop instilled into each eye (OU), 4 times daily (QID), approximately 4 hours apart
  Arms: Brimonidine tartrate ophthalmic solution 0.025% with sodium hyaluronate (BTOS-HA)
Drug: Lumify® — Brimonidine tartrate ophthalmic solution 0.025%, administered as 1 topical ocular drop instilled into each eye (OU), 4 times daily (QID), approximately 4 hours apart
  Arms: Brimonidine tartrate ophthalmic solution 0.025%

SUMMARY:
To demonstrate the efficacy of BTOS-HA as non inferior to Lumify for treating ocular redness in a population of adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily provide written informed consent
2. ≥18 years of age
3. Able and willing to follow instructions, including participation in all trial assessments and visits
4. History of vasoconstrictor (redness relief drops) use within the last 6 months, or a desire to use over the counter (OTC) vasoconstrictors for redness relief
5. Able to self-administer eye drops satisfactorily
6. A calculated best-corrected (if necessary) visual acuity of 0.3 logarithm of the minimum angle of resolution (logMAR) or better in each eye, as measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart
7. Show a baseline redness score >1 in both eyes as scored by the investigator using the Investigator Ocular Redness Scale (range 0-4)
8. Stable ocular health at Visit 2 (Day 1), (defined as no ocular conditions requiring therapy or surgical intervention during the study).

Exclusion Criteria:

1. Known contraindications or sensitivity to the use of any of the investigational drug(s) or their components, or any other medications required by the protocol
2. Ocular surgery within 3 months prior to screening and/or a history of refractive surgery within the past 6 months, and/ or planned surgery (ocular or systemic) during the trial period or within 30 days after the study period
3. Have the presence of an active ocular infection (bacterial, viral, or fungal) or positive history of an ocular herpetic infection
4. Use any of the following disallowed medications during the period indicated prior to randomization or planned use during the study:

   1. All topical ophthalmic agents including artificial tear products, eye whiteners (e.g., vasoconstrictors), ocular decongestants, ocular antihistamines, ocular corticosteroids, dilating drops (excluding dilated ophthalmoscopy exam at Visit 2), and contact lenses: 5 days
   2. Systemic antihistamines or decongestants: 7 days
   3. Systemic corticosteroids or cancer chemotherapy, and/or any other systemic medications which the investigator feels may confound study data, put the subject at risk or interfere with subject's study participation: 14 days
5. Have prior (within 7 days of beginning investigational drug) or currently active significant illness that could compromise participation, in the opinion of the investigator
6. Have prior (within 30 days of beginning investigational drug) or anticipated concurrent use of an investigational drug or device during the study period
7. Have an ocular or systemic condition or a situation which, in the investigator's opinion, may put the subject at increased risk, confound study data, or interfere significantly with the subject's study participation (e.g., blepharitis, active ocular allergies, rosacea with peri-ocular involvement, uncontrolled diabetes, hypertension, or cardiovascular disease).
8. Have a diagnosis of ocular hypertension or glaucoma at screening
9. Any female who is nursing, lactating, pregnant, planning a pregnancy, or has a positive urine pregnancy test at Visit 2 (Day 1).
10. Any female of childbearing potential (FOCBP) who is unwilling to: a) agree to have urine pregnancy testing performed at Visit 2 (Day 1), and b) agree to use at least 1 medically acceptable form of birth control for at least 14 days prior to the first dose of study drug at Visit 2 (Day 1), throughout the study duration, and for 1 month after the last dose of investigational drug at Visit 4 (Day 29) NOTE: FOCBP include all females who have experienced menarche and have not experienced menopause (as defined by amenorrhea for greater than 12 consecutive months) or have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy)

    NOTE: Acceptable forms of birth control include:
    * Mechanical (spermicide in conjunction with a barrier such as a diaphragm or condom)
    * Hormonal contraceptive (oral, injectable, implantable, or transdermal)
    * Intrauterine device, or
    * Surgical sterilization of male partner at least 3 months prior to the first dose of investigational drug at Visit 2 (Day 1)

    NOTE: For non-sexually active female subjects, abstinence may be regarded as an adequate method of birth control when this is in line with the preferred and usual lifestyle of the subject; however, if the subject becomes sexually active during the trial, she must agree to use adequate birth control as defined above for the remainder of the trial
11. Any male who is unwilling to agree to use at least 1 medically acceptable form of birth control with female partner (FOCBP)

NOTE: Acceptable forms of birth control include:

* True abstinence (when this is in line with the preferred and usual lifestyle of the subject), or
* Vasectomy at least 3 months prior to the first dose of study drug at Visit 2 (Day 1)

Without a vasectomy, must use condoms with spermicidal foam/gel/film/cream/suppository at least 14 days prior to the first dose of investigational drug at Visit 2 (Day 1) and throughout the study duration, and for 1 month after the last dose of the investigational drug at Visit 4 (Day 29)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 578 (Actual)
Dates: Start 2025-05-22 (Actual); Primary Completion 2025-06-29 (Actual); Study Completion 2025-06-29 (Actual)

PRIMARY OUTCOMES:
Ocular redness score (0-4 unit scale, allowing half-unit increments) evaluated by the investigator at Visit 2 (Day 1) | Assessed at Visit 2 (Day 1) prior to investigational drug instillation and after investigational drug instillation at 5(+1) minutes, 15(+1) minutes, 30(+1) minutes, 60(+10) minutes, 90(+10) minutes, 120(+15) minutes, 180(+15) minutes, 240(+15) minutes
  Ocular redness score (0-4 unit scale, allowing half-unit increments) evaluated by the investigator at Visit 2 (Day 1) prior to investigational drug instillation and after investigational drug instillation at 5(+1) minutes, 15(+1) minutes, 30(+1) minutes, 60(+10) minutes, 90(+10) minutes, 120(+15) minutes, 180(+15) minutes, 240(+15) minutes

SECONDARY OUTCOMES:
Change from pre-instillation ocular redness score (0-4 unit scale, allowing half-unit increments) evaluated by the investigator at Visit 2 (Day 1) | Assessed at Visit 2 (Day 1) after investigational drug instillation evaluated hierarchically at: 1 (+0.5) minute, 360 (+15) minutes and 480 (+15) minutes
  Change from pre-instillation ocular redness score (0-4 unit scale, allowing half-unit increments) evaluated by the investigator at Visit 2 (Day 1) after investigational drug instillation evaluated hierarchically at: 1 (+0.5) minute, 360 (+15) minutes and 480 (+15) minutes
Change from pre-instillation ocular redness score (0-4 unit scale, allowing half-unit increments) evaluated by the Investigator after investigational drug instillation evaluated hierarchically at Visit 3 (Day 15) | Assessed at Visit 3 (Day 15) 5 (+1) minutes and 15 (+1) minutes
  Change from pre-instillation ocular redness score (0-4 unit scale, allowing half-unit increments) evaluated by the Investigator after investigational drug instillation evaluated hierarchically at Visit 3 (Day 15) 5 (+1) minutes and 15 (+1) minutes
Change from pre-instillation ocular redness score (0-4 unit scale, allowing half-unit increments) evaluated by the Investigator after investigational drug instillation evaluated hierarchically at Visit 4 (Day 29) | Assessed at Visit 4 (Day 29) 5 (+1) minutes and 15 (+1) minutes
  Change from pre-instillation ocular redness score (0-4 unit scale, allowing half-unit increments) evaluated by the Investigator after investigational drug instillation evaluated hierarchically at Visit 4 (Day 29) 5 (+1) minutes and 15 (+1) minutes
Change from pre-instillation ocular redness score (0-4 unit scale, allowing half-unit increments) evaluated by the investigator after investigational drug instillation at Visit 2 (Day 1) | Assessed at Visit 2 (Day 1) evaluated hierarchically at 0.5 (+0.25) minute and 600 (+15) minutes
  Change from pre-instillation ocular redness score (0-4 unit scale, allowing half-unit increments) evaluated by the investigator after investigational drug instillation at Visit 2 (Day 1) evaluated hierarchically at 0.5 (+0.25) minute and 600 (+15) minutes

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Site 102, Glendale, California
  - Site 104, Newport Beach, California
  - Site 111, Northbrook, Illinois
  - Site 109, Pittsburg, Kansas
  - Site 106, Louisville, Kentucky
  - Site 103, Andover, Massachusetts
  - Site 108, Garner, North Carolina
  - Site 107, Shelby, North Carolina
  - Site 112, Cranberry Township, Pennsylvania
  - Site 101, Memphis, Tennessee
  - Site 105, Smyrna, Tennessee

IPD SHARING:
Plan to Share IPD: No